CLINICAL TRIAL: NCT03383289
Title: Resident-to-Resident Elder Mistreatment Intervention for Dementia Care in Assisted Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew Home at Riverdale (Other)
Collaborators: Cornell University (Other); Weill Medical College of Cornell University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 952; 5R01AG057389 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-26 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Assisted Living, Resident to Resident Elder Mistreatment

STUDY DESIGN:
Who Masked: Participant
Masking Description: Research Assistants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-REM training (Experimental): 3 module training for frontline staff in assisted living facilities related to recognizing and management of resident-to-resident elder mistreatment
  Interventions: Other: R-REM training
- Usual Care (No Intervention): Usual care arm

INTERVENTIONS:
Other: R-REM training — three training modules for front-line long-term care staff to aid in recognition, management and reporting of R-REM
  Arms: R-REM training

SUMMARY:
Resident-to-resident elder mistreatment (R-REM) is a significant problem in long-term services and support settings (LTSS), and likely to cause physical and or psychological distress. The proposed project tests an intervention developed for use by LTSS staff. As such, it represents an important step in the process of developing approaches for ameliorating and preventing R-REM in assisted living residences which house residents with dementia and related behavioral disorders, and is thus likely to have significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* all long term residents residing at each facility at baseline, for those unable to consent, proxy consent will be sought

Exclusion Criteria:

* residents receiving hospice care,
* facilities will have the option to exclude individuals for selected reasons, (e.g., severe psychosis)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 930 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne A Teresi, PhD, EdD, Principal Investigator — Research Division, Hebrew Home at Riverdale
Locations (1):
- Hebrew Home at Riverdale, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teresi JA, Silver S, Boratgis GD, Schultz L, Meador R, Kong J, Eimicke JP, Lachs MS, Pillemer KA. A Staff Intervention Targeting Resident-to-Resident Aggression in Assisted Living: A Cluster-Randomized Trial. J Am Geriatr Soc. 2026 Jan 9. doi: 10.1111/jgs.70268. Online ahead of print. PMID 41511825
- [Derived] Teresi JA, Silver S, Ramirez M, Kong J, Eimicke JP, Boratgis GD, Meador R, Schultz L, Lachs MS, Pillemer KA. Resident-to-resident elder mistreatment (R-REM) intervention for direct care staff in assisted living residences: study protocol for a cluster randomized controlled trial. Trials. 2020 Aug 12;21(1):710. doi: 10.1186/s13063-020-04580-z. PMID 32787944

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Assisted Living Facilities
Groups:
- R-REM Training to Improve Recognition and Reporting: 3 module training for frontline staff in assisted living facilities related to recognizing and management of resident-to-resident elder mistreatment, including the Support, Evaluate, Act, Report, Care plan, and Help to avoid (SEARCH) approach
Period: Overall Study
Arm/Group | R-REM Training to Improve Recognition and Reporting | Usual Care
Started | 495; 7 Assisted Living Facilities | 435; 7 Assisted Living Facilities
Study Completion (Given intent-to-treat design, all those enrolled are considered to have completed the study) | 495; 7 Assisted Living Facilities | 435; 7 Assisted Living Facilities
Completed | 324; 7 Assisted Living Facilities | 272; 7 Assisted Living Facilities
Not Completed | 171; 0 Assisted Living Facilities | 163; 0 Assisted Living Facilities
Not completed — Death | 83 | 78
Not completed — discharge from facility | 84 | 84
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- R-REM Training Intervention to Improve Recognition and Reporting: 3 module training for frontline staff in assisted living facilities related to recognizing and management of resident-to-resident elder mistreatment, including the Support, Evaluate, Act, Report, Care plan, and Help to avoid (SEARCH) approach
- Usual Care: Usual care arm. Assisted Living facilities assigned to Usual Care.
- Total: Total of all reporting groups
Arm/Group | R-REM Training Intervention to Improve Recognition and Reporting | Usual Care | Total
Number analyzed (Participants) | 495 | 435 | 930
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 990 is not the correct total number of participants. It is 930.
  years | 87.68 (6.92) | 88.36 (7.52) | 88.00 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 990 is not the correct total number of participants. The total number of participants is 930.
  Participants
    Female | 392 | 346 | 738
    Male | 103 | 89 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 990 is not the correct total number of participants. The correct total number of participants is 930.
  Participants
    Hispanic or Latino | 2 | 7 | 9
    Not Hispanic or Latino | 363 | 320 | 683
    Unknown or Not Reported | 130 | 108 | 238
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 8 | 11
  White | 476 | 418 | 894
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 2 | 13
Region of Enrollment [Number; unit: Participant] — Population: 990 is not the correct total number of participants. The total number of participants is 930.
  Participant
    United States | 495 | 435 | 930

OUTCOME MEASURES:

1. Primary Outcome: Falls, Accidents, and Injuries
Description: Impact on falls, accidents, and injuries as measured by incident reports
Time Frame: Six months before baseline through twelve month follow-up
Population: Analyses were intent to treat. All those randomized were included.
Measure: Number; unit: participants
Arm/Group | R-REM Training to Improve Recognition and Reporting | Usual Care
Number analyzed (Participants) | 495 | 435
participants | 141 | 115
Statistical Analysis 1: Comparison: R-REM Training to Improve Recognition and Reporting vs Usual Care; Test type: Superiority; p = 0.4170, Mixed Models Analysis; MIANALYZE was used to model missing data. Models were adjusted for the design effects of clustering; Beta estimate of the percent who fell = 0.118, Standard Error of Mean 0.145

2. Secondary Outcome: Affect
Description: Impact on participant affect as measured by the Feeling Tone Questionnaire (FTQ). A 16-item scale with a theoretical range of 0-32. Higher score indicates lower affect (depressed direction).
Time Frame: Baseline, 6- and 12- month follow-up
Population: The FTQ was collected only on the subset of participants who were capable of response
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-REM Training Intervention to Improve Recognition and Reporting | Usual Care
Number analyzed (Participants) | 279 | 259
score on a scale
  Baseline | 6.29 (5.16) | 6.65 (4.79)
  6-month follow up | 6.37 (5.92) | 6.44 (4.95)
  12-month follow-up | 5.30 (4.10) | 6.11 (4.47)

3. Other Pre Specified Outcome: Staff Knowledge Module 1
Description: Module 1: Recognizing R-REM 10-item knowledge test related to recognizing resident-to-resident elder mistreatment The potential (theoretical) total score range is 0-10 with a higher score indicating more knowledge (better outcome)
Time Frame: Pre and post training evaluation: Immediately before and immediately after training
Population: Front-line staff in Intervention group nursing homes. Please note that this n differs from the participant n (assisted living residents) described in the flow diagram because this outcome is based on a different sample (staff).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- R-REM Training to Improve Recognition and Reporting - Immediate Pretest: 3 module training for frontline staff in assisted living facilities related to recognizing and management of resident-to-resident elder mistreatment including the Support, Evaluate, Act, Report, Care plan, and Help to avoid (SEARCH) approach Note: Knowledge tests were only given to staff in Intervention sites. No knowledge tests were obtained in usual care facilities.
- R-REM Training to Improve Recognition and Reporting - Immediate Posttest: Knowledge test scores administered immediately after the training was provided Note: Knowledge tests were only given to staff in Intervention sites. No knowledge tests were obtained in usual care facilities.
Arm/Group | R-REM Training to Improve Recognition and Reporting - Immediate Pretest | R-REM Training to Improve Recognition and Reporting - Immediate Posttest
Number analyzed (Participants) | 211 | 211
score on a scale | 6.17 (1.97) | 7.53 (1.95)
Statistical Analysis 1: Comparison: R-REM Training to Improve Recognition and Reporting - Immediate Pretest vs R-REM Training to Improve Recognition and Reporting - Immediate Posttest; Analysis of adjusted mean differences using a paired t test procedure; Test type: Other — paired t test; p < 0.001, paired t test; Mean Difference (Final Values) = -1.353, 95% CI 2-sided [-1.708 to -0.998], Standard Error of Mean 0.181

4. Other Pre Specified Outcome: Staff Recognition, Reporting and Care Planning of Resident-to-resident Elder Mistreatment Events
Description: Statistical Analysis 1: Count of participants with events reported by the staff through the informant interview measure Statistical Analysis 2: Count of events reported through the Behavior Recognition Documentation Sheets (BRDS)
Time Frame: baseline through 1-year follow-up
Population: Nursing home staff informants.
Measure: Count of Participants; unit: Participants
Arm/Group | R-REM Training to Improve Recognition and Reporting | Usual Care
Number analyzed (Participants) | 478 | 415
Participants | 478 | 415
Statistical Analysis 1: Comparison: R-REM Training to Improve Recognition and Reporting vs Usual Care; Test type: Superiority; p = 0.0064, Poisson regression; Beta = 0.6364, 95% CI 2-sided [0.1797 to 1.0931], Standard Error of Mean 0.2330
Statistical Analysis 2: Comparison: R-REM Training to Improve Recognition and Reporting vs Usual Care; Test type: Superiority; p = 0.001, Poisson regression; Estimated log mean = -4.0168, 95% CI 2-sided [-5.5827 to -2.4509]

5. Other Pre Specified Outcome: Staff Knowledge Module 2
Description: Module 2: Management of R-REM 10-item knowledge tests The potential (theoretical) range is 0-10 with a higher score indicating more knowledge (better outcome)
Time Frame: Administered immediately before and immediately after training was provided
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- R-REM Training to Improve Recognition and Reporting Pre-test: 3 module training for frontline staff in assisted living facilities related to recognizing and management of resident-to-resident elder mistreatment including the Support, Evaluate, Act, Report, Care plan, and Help to avoid (SEARCH) approach administered immediately before training provided
- R-REM Training to Improve Recognition and Reporting Post-test: Knowledge test scores immediately post training Note: Knowledge tests were only given to staff in intervention sites. No knowledge tests were obtained in usual care facilities.
Arm/Group | R-REM Training to Improve Recognition and Reporting Pre-test | R-REM Training to Improve Recognition and Reporting Post-test
Number analyzed (Participants) | 228 | 228
score on a scale | 7.59 (2.00) | 8.04 (1.52)
Statistical Analysis 1: Comparison: R-REM Training to Improve Recognition and Reporting Pre-test vs R-REM Training to Improve Recognition and Reporting Post-test; Test type: Other — adjusted mean differences from paired t tests; p = 0.005, paired t test; Mean Difference (Final Values) = -0.456, 95% CI 2-sided [-0.774 to -0.138], Standard Error of Mean 0.162

ADVERSE EVENTS:
Time Frame: 1 year
Description: Using the definitions from clinicaltrials.gov, the DSMB reviewed all events
Arm/Group | R-REM Training | Usual Care
All-Cause Mortality (participants affected / at risk) | 83/495 | 78/435
Serious Adverse Events (participants affected / at risk) | 0/495 | 0/435
Other Adverse Events (participants affected / at risk) | 0/495 | 0/435

LIMITATIONS AND CAVEATS:
The pandemic may have affected the observed affect and behavior results which may have been impacted by missing data. During the pandemic there was more social isolation, impacting quality-of-life outcomes. There were several limitations to this study, most notably the large amount of missing data observed at the final wave in part because of COVID, affected testing the third study aim. To mitigate this loss, several statistical methods were used to examine missing data due to COVID.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT03383289/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT03383289/ICF_001.pdf